CLINICAL TRIAL: NCT03032731
Title: Trial of a Self-directed Behaviour Change Intervention for Physical Activity and Healthy Eating.
Brief Title: Trial of a New Online Programme for Physical Activity and Healthy Eating.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Elisabeth Grey, Principal investigator, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EP 16/17 034
Record Dates: First submitted 2017-01-19; First posted 2017-01-26 (Estimated); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Overweight/Obesity
Keywords: Physical activity; Diet; Health Behavior
MeSH Terms: conditions — Overweight; Obesity; Motor Activity; Health Behavior

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Website and pedometer Intervention (Experimental): Participants allocated to this group will be given a one-off set-up session in which a researcher will show them the intervention website, create a user profile for them and provide guidance on how to use the site to gain health information, set personal behavioural goals and record and monitor their behaviour in relation to their goals. The researcher will also provide the participant with a pedometer and instruct them how to use this and where they can record their daily steps on the website. For 6 weeks, participants will be asked to use the website and be sent weekly email reminders to do so and log their goal progress. After 6 weeks, no further emails will be sent but participants will still be able to access the website and use the pedometer if they wish.
  Interventions: Behavioral: Website and pedometer intervention
- Control (Other): Participants allocated to this group will be given a one-off session in which a researcher shows them publicly available web-based resources for health behaviour change (provided by the National Health Service (NHS)). Like those participants in the intervention group, they will be assessed again after 6 and 12 weeks. Participants in the control arm will be offered the intervention (access to the study website and a pedometer) after 12 weeks.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Website and pedometer intervention — Self-directed, website-based intervention delivered with a pedometer to promote understanding of health and health behaviour change.
  Arms: Website and pedometer Intervention
Other: Control — Standard, publicly available NHS resources for healthy lifestyles.
  Arms: Control

SUMMARY:
Many healthy lifestyle interventions have been developed to help people change their activity and diet, lose weight and thus reduce their risk of developing type 2 diabetes (T2DM) and cardiovascular disorders (CVD). However, these interventions often fail to engage their target audience, which undermines their effectiveness in changing behaviour and health outcomes.

The purpose of this study is to investigate the effectiveness of a self-directed, website-based intervention to promote physical activity and healthy dietary behaviours. The intervention frames health information from a novel perspective, which our previous work has indicated can help to promote interest in the health information and improve attitudes, self-efficacy and motivation towards physical activity and healthy dietary behaviours.

The intervention comprises a website of information resources and personal recording areas to set goals and monitor activity and diet, weekly emails and pedometers. In this trial we aim to see whether the intervention has any impact on people's physical activity and diet, as well as their risk of developing CVD and T2DM. The intervention will be compared with a control condition in which participants will be shown standard resources available on NHS websites. Overweight/obese (BMI 25 - 39.5) males and females aged 35-74 years will be recruited from the community. The active intervention will last 6 weeks (during this period participants will receive weekly emails from the research team) and there will be a 6-week follow-up phase (in which participants will still have access to the website but contact from the research team). Activity, diet, disease risk markers and psychological antecedents of behaviour will be assessed at baseline, post-intervention (6-weeks) and post follow-up (12- weeks).

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent to participate in the study.
* Male or female and aged between 35-74 years.
* Defined as overweight or obese, i.e. BMI>25kg/m2.
* Able to travel to the university for assessment days.

Exclusion Criteria:

* Individuals who are not fluent in the English language, and who do not have access to and do not regularly use the internet and an email account.
* Individuals diagnosed with coronary heart disease, chronic kidney disease, type 2 diabetes, stroke, heart failure, severe hypertension (BP>180/110mmHg) and peripheral arterial disease.
* BMI>40kg/m2 (morbidly obese).
* Currently using weight loss drugs or other medication that can affect weight.
* Any reported recent (i.e. last 6 months) shift (>5%) in body mass or large change in habitual lifestyle.
* Individuals unable to change their physical activity (e.g. through disability).
* Current (pre-baseline) or recent (i.e. last 2 months) participation in another research trial or lifestyle supportive intervention or referral.
* Pregnant

Ages: 35 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2017-09-12 (Actual); Study Completion 2017-09-12 (Actual)

PRIMARY OUTCOMES:
Change in mean daily physical activity level (PAL) | Baseline, 6 weeks and 12 weeks after starting the intervention/control period
  Mean daily physical activity level (PAL) will be assessed using accelerometers (BodyMedia, worn on the upper arm), worn for a continuous 7-day period, being removed during this time only for water-based activities such as showering or swimming. The accelerometers gather minute by minute total energy expenditure (TEE) data, which will be used to calculate PAL (PAL = TEE/BMR, where BMR = basal metabolic rate, to be calculated using the Schofield equation).
Change in mean daily energy intake (EI) | Baseline, 6 weeks and 12 weeks after starting the intervention/control period
  Mean daily energy intake (EI) will be assessed using 3-day weighed food diaries, incorporating 2 week days and 1 weekend day .

SECONDARY OUTCOMES:
Fasting plasma glucose concentration | Baseline, 6 weeks and 12 weeks after starting the intervention/control period
  Comparison of glucose concentration in the blood plasma at rest across all three measurement points.
Fasting plasma insulin concentration | Baseline, 6 weeks and 12 weeks after starting the intervention/control period
  Comparison of insulin concentration in the blood plasma at rest across all three measurement points.
Fasting triglyceride concentration | Baseline, 6 weeks and 12 weeks after starting the intervention/control period
  Comparison of triglyceride concentration in the blood serum at rest across all three measurement points.
Fasting total cholesterol concentration | Baseline, 6 weeks and 12 weeks after starting the intervention/control period
  Comparison of total concentration in the blood serum at rest across all three measurement points.
Fasting LDL cholesterol concentration | Baseline, 6 weeks and 12 weeks after starting the intervention/control period
  Comparison of LDL concentration in the blood serum at rest across all three measurement points.
Fasting HDL cholesterol concentration | Baseline, 6 weeks and 12 weeks after starting the intervention/control period
  Comparison of HDL concentration in the blood serum at rest across all three measurement points.
C-reactive protein (CRP) concentration | Baseline, 6 weeks and 12 weeks after starting the intervention/control period
  Comparison of CRP concentration in the blood serum at rest across all three measurement points.
Body mass index (BMI) | Baseline, 6 weeks and 12 weeks after starting the intervention/control period
  Comparison of BMI (defined as mass in kg divided by height in metres squared) across all three measurement points.
Waist circumference | Baseline, 6 weeks and 12 weeks after starting the intervention/control period
  Comparison of waist circumference (in centimetres) across all three measurement points.
Blood pressure | Baseline, 6 weeks and 12 weeks after starting the intervention/control period
  Comparison of blood pressure (systolic/diastolic mmHG) across all three measurement points.
Quality of diet | Baseline, 6 weeks and 12 weeks after starting the intervention/control period
  Diet quality will be assessed based on the proportion of fibre, free sugars and refined carbohydrates, and saturated fats in the diet. The intervention aims to promote an increase in fibre intake and decrease in free sugar, refined carbohydrate and saturated fat intake. Data will be collected using 3-day weighed food diaries, incorporating 2 week days and 1 weekend day.
Motivation for physical activity | Baseline, 6 weeks and 12 weeks after starting the intervention/control period
  Motivation will be assessed using the Behavioural Regulation for Exercise Questionnaire 3 (BREQ 3: Markland & Tobin, 2004; Wilson, Rodgers, Loitz & Scime, 2006) adapted for physical activity.
Motivation for healthy eating | Baseline, 6 weeks and 12 weeks after starting the intervention/control period
  Motivation will be assessed using the Behavioural Regulation for Exercise Questionnaire 3 (BREQ 3: Markland & Tobin, 2004; Wilson, Rodgers, Loitz & Scime, 2006) adapted for diet.
Self-efficacy for physical activity and healthy eating | Baseline, 6 weeks and 12 weeks after starting the intervention/control period
  Self-efficacy will be measured using the Barriers Self-Efficacy Scale for Exercise (BARSE; McAuley, 1992) adapted for physical activity.
Self-efficacy for healthy eating | Baseline, 6 weeks and 12 weeks after starting the intervention/control period
  Self-efficacy will be measured using the self-efficacy scale for eating a healthy diet developed by Pawlak and Colby (2009).

CONTACTS AND LOCATIONS:
Overall Officials: Dylan Thompson, PhD, Principal Investigator — University of Bath
Locations (1):
- University of Bath, Bath, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grey EB, Thompson D, Gillison FB. Effects of a Web-Based, Evolutionary Mismatch-Framed Intervention Targeting Physical Activity and Diet: a Randomised Controlled Trial. Int J Behav Med. 2019 Dec;26(6):645-657. doi: 10.1007/s12529-019-09821-3. PMID 31654276